CLINICAL TRIAL: NCT07156201
Title: A First-in-Human, Phase 1a, Randomized, Double-Blinded, Placebo-Controlled, Single- and Multiple-Ascending Dose and Food Effect Study to Assess the Safety, Tolerability, and Pharmacokinetics of ABS-1230 Administered Orally to Healthy Adults
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of ABS-1230 Given Orally Compared With Placebo in Healthy Participants Aged 18 to 55 Years
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Actio Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABS1230-1001
Record Dates: First submitted 2025-08-25; First posted 2025-09-05 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: KCNT1-Related Epilepsy
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- ABS-1230 Single Dose (Experimental): Single doses of ABS-1230
  Interventions: Drug: ABS-1230
- ABS-1230 Multiple Doses (Experimental): Multiple doses of ABS-1230
  Interventions: Drug: ABS-1230
- Placebo Single Dose (Placebo Comparator): Single doses of placebo
  Interventions: Drug: Placebo
- Placebo Multiple Doses (Placebo Comparator): Multiple doses of placebo
  Interventions: Drug: Placebo
- ABS-1230 Singe Dose + Omeprazole (Experimental): Single doses of ABS-1230 + omeprazole
  Interventions: Drug: ABS-1230; Drug: Omeprazole

INTERVENTIONS:
Drug: ABS-1230 — ABS-1230
  Arms: ABS-1230 Multiple Doses; ABS-1230 Singe Dose + Omeprazole; ABS-1230 Single Dose
Drug: Placebo — Placebo
  Arms: Placebo Multiple Doses; Placebo Single Dose
Drug: Omeprazole — Omeprazole
  Arms: ABS-1230 Singe Dose + Omeprazole

SUMMARY:
This first in human trial will evaluate the safety, tolerability, and pharmacokinetics of single ascending doses, multiple ascending doses, and fed and fasted doses of ABS-1230 given orally compared with placebo in adult healthy participants.

DETAILED DESCRIPTION:
This is a Phase 1a, first-in-human, placebo-controlled study consisting of 3 parts.

Part 1 is a single ascending dose (SAD) study in up to 32 participants consisting of a screening period of up to 28 days prior to a single dose of ABS-1230 or placebo, with follow-up 7 days and 14 days after dosing.

Part 2 is a multiple ascending dose (MAD) study in up to 30 participants consisting of a screening period of up to 28 days, followed by ABS-1230 or placebo once daily for 14 days, with follow-up 7 days and 14 days after dosing is completed.

Part 3 is a food effect (FE) study in 12 participants consisting of two doses of ABS-1230 under fasted and fed conditions and in combination with omeprazole with follow-up 7 days and 14 days after dosing is completed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 55 years, inclusive
* Body mass index greater than or equal to 18 to less than or equal to 32 kg/m2
* Medically healthy with no clinically significant medical history, physical examination, vital sign, standard 12-lead ECG, chemistry, hematology, urinalysis, or coagulation results at Screening as deemed by the Investigator
* Male and female subjects must use adequate birth control and agree not to donate sperm or eggs for the time periods specified in the protocol

Exclusion Criteria:

* Positive result for HIV, HBV, or HCV
* History of malignancy other than treated basal cell carcinoma, squamous cell carcinoma, or carcinoma in situ of the cervix
* History of alcoholism or recreational drug use within 2 years or a positive alcohol or tobacco test result at screening or first check-in visit
* For female participants, must not be pregnant, breastfeeding, or seeking to become pregnant while in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability (incidence, severity, and dose-relationship of adverse events) | Measured from Day 1 to End of Study or Early Termination (up to 4 weeks)
  To assess safety and tolerability of ABS-1230 following single and multiple oral administration by determining the incidence, severity, and dose-relationship of adverse events
Safety and tolerability (incidence, severity, and dose-relationship of clinically significant changes in laboratory parameters) | Measured from Day 1 to End of Study or Early Termination (up to 4 weeks)
  To assess safety and tolerability of ABS-1230 following single and multiple oral administration by determining the incidence, severity, and dose-relationship of clinically significant laboratory changes

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] After Single Dose of ABS-1230 | Measured from Day 1 to End of Study or Early Termination (up to 2 weeks)
  To evaluate the pharmacokinetics of single dose of ABS-1230
Maximum Plasma Concentration [AUCtau] After Single Dose of ABS-1230 | Measured from Day 1 to End of Study or Early Termination (up to 2 weeks)
  To evaluate the pharmacokinetics of single dose of ABS-1230
Maximum Plasma Concentration [Cmax] After Multiple Doses of ABS-1230 | Measured from Day 1 to End of Study or Early Termination (up to 4 weeks)
  To evaluate the pharmacokinetics of multiple doses of ABS-1230
Maximum Plasma Concentration [AUCtau] After Multiple Doses of ABS-1230 | Measured from Day 1 to End of Study or Early Termination (up to 4 weeks)
  To evaluate the pharmacokinetics of multiple doses of ABS-1230
Maximum Plasma Concentration [Cmax] After Fed, Fasted and in Combination with Omeprazole Doses of ABS-1230 | Measured from Day 1 to End of Study or Early Termination (up to 4 weeks)
  To evaluate the pharmacokinetics of fed, fasted, and in combination with omeprazole doses of ABS-1230
Maximum Plasma Concentration [AUCtau] After Fed, Fasted and in Combination with Omeprazole Doses of ABS-1230 | Measured from Day 1 to End of Study or Early Termination (up to 4 weeks)
  To evaluate the pharmacokinetics of fed, fasted, and in combination with omeprazole doses of ABS-1230

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Actio Bioscences, Inc.
Locations (1):
- Scientia Clinical Research, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No